CLINICAL TRIAL: NCT05329844
Title: Randomized, Open Label, Two-sequence, Two-treatment, Two-period, Crossover, Single Dose Bioequivalence Study of Vildagliptin Tablets 50 mg of AET Laboratories Pvt. Ltd., India With Galvus 50 mg Tablets of Novartis Europharm Ltd., United Kingdom in Normal Healthy, Adult, Male Human Subjects Under Fasting Conditions.
Brief Title: The Study Aims to Show Bioequivalence of the Test Product and the Reference Reference Product in a Crossover Design Study Healthy Volunteers. Additionally, the Safeyt Profile of Test Product Compared to Reference Product Will be Assessed.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AET Laboratories Private Limited (Industry)
Responsible Party: Sponsor
Organization: Alfred E. Tiefenbacher (GmbH & Co. KG) (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 13-VIN-343
Record Dates: First submitted 2022-03-25; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vildagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vildagliptin 50 mg Tablet (Experimental): 1 tablet of Vildagliptin 50 mg as single-dose administration
  Interventions: Drug: Vildagliptin 50 MG
- Galvus 50 mg Tablet (Active Comparator): 1 tablet of Galvus 50 mg (each tablet contains 50 mg Vildagliptin) as single-dose administration
  Interventions: Drug: Vildagliptin 50 MG

INTERVENTIONS:
Drug: Vildagliptin 50 MG — 50 mg Vildagliptin as single-dose per study period

SUMMARY:
To evaluate and compare the relative bioavailability and therefore the bioequivalence of Vildagliptin Tablets 50 mg of AET Laboratories Private Limited, India, with GALVUS® 50 mg Tablets of Novartis Europharm Limited, United Kingdom, in normal, healthy, adult, male human subjects under fasting conditions and to evaluate the safety and tolerability of Vildagliptin Tablets 50 mg in normal, healthy, adult, male human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged between 18 and 45 years (both inclusive).
2. Subjects' weight within the normal range according to normal values for the Body Mass Index (18.5 to 30 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within clinically acceptable normal range.
4. Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
5. Subjects having clinically acceptable chest X-Ray.
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine and morphine).
7. Subjects having negative alcohol breath test.
8. Subjects willing to adhere to the protocol requirements and to provide written informed consent.
9. No history or presence of smoking.
10. No history or presence of alcoholism and drug of abuse.

Exclusion Criteria:

1. Hypersensitivity to Vildagliptin or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month of the study starting.
4. History or presence of asthma, urticaria or other significant allergic reactions.
5. History or presence of significant gastric and/or duodenal ulceration.
6. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
7. History or presence of cancer.
8. Difficulty with donating blood.
9. Difficulty in swallowing solids like tablets or capsules.
10. Use of any prescribed or OTC medication during last two weeks prior to Dosing in Period 01.
11. Major illness during 3 months before screening.
12. Participation in a drug research study within past 3 months.
13. Donation of blood in the past 3 months before screening.
14. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
15. History or presence of significant easy bruising or bleeding.
16. History or presence of significant recent trauma.
17. Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cmax of Vildagliptin for the test and reference products | up to 24 hours
  The maximum concentration in plasma among observed concentrations at pre-specified time points
AUC0-t of Vildagliptin for the test and the reference products | up to 24 hours
  The area under the plasma concentration versus time curve from time 0 to the last measured concentration

SECONDARY OUTCOMES:
AUC0-∞ of Vildagliptin for the test and the reference products | up to 24 hours
  The area under the plasma concentration versus time curve from time 0 to to infinite time
Tmax of Vildagliptin for the test and the reference products | up to 24 hours
  The time to maximum measured plasma concentration
T1/2 of Vildagliptin for the test and the reference products | up to 24 hours
  Plasma elimination half-life
Kel of Vildagliptin for the test and the reference products | up to 24 hours
  Elimination rate constant
Number of treatment-related adverse events (AE) for the test and the reference products as assessed by guidance predefined in the protocol | through study completion, an average of 1 month
  An AE is defined as any untoward medical occurrence in a subject administered the test or the reference product and which does not necessarily have a causal relationship with the treatment.